CLINICAL TRIAL: NCT00186264
Title: Does Concurrent Hydrocortisone With Venlafaxine XR Speed Antidepressant Response?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Principal Investigator, Charles DeBattista, Professor of Psychiatry and Behavioral Sciences, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Wyeth 0600B-100625
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2019-10-04 (Actual); Status verified 2019-10

CONDITIONS: Depressive Disorder, Major
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Hydrocortisone

INTERVENTIONS:
Drug: venlafaxine XR
Drug: hydrocortisone

SUMMARY:
The primary purpose of this study is to examine whether IV hydrocortisone can speed up the time required for Venlafaxine XR to work.

DETAILED DESCRIPTION:
Participants will be treated with Venlafaxine XR for 6 weeks. The dose of Venlafaxine XR will begin at 37.5 mg/day and be gradually increased to a maximum of 225 mg/day. The dose may be kept as low as 75 mg/day if necessary. Study doctor will be assessing mood to determine if some patients respond more quickly than the several weeks often required for an antidepressant to begin working. On the first day of treatment with Venlafaxine XR, participant will be randomly assigned (similar to a flip of a coin) to receive hydrocortisone 15 mg /day or placebo for two days. Placebo is an inactive substance, like a sugar pill. This dose of hydrocortisone is less than a typical replacement dose for patients who are not producing cortisol (hydrocortisone) naturally. The hydrocortisone is administered intravenously (in a vein) over the course of 2 hours for two consecutive days. Neither participant nor study doctor will know which treatment participant is receiving. However, this information is available to study doctor if it is needed.

ELIGIBILITY:
Inclusion Criteria::- outpatients at least 18 years of age

* current major depressive episode
* HDRS greater than or equal to 21
* good physical health Exclusion Criteria:- history of sensitivity, intolerance, or non-response to venlafaxine
* history of sensitivity to hydrocortisone
* history of bipolar 1 illness
* meets DSM-IV criteria for a current or past psychotic disorder
* meets DSM-IV criteria for substance abuse or dependence in previous 6 months
* significant imminent suicide risk
* medical condition that would compromise participation in the study
* woman of child bearing potential not using adequate birth control in the opinion of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2002-08 (Actual); Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
To determine if treatment of major depression with hydrocortisone concurrent with starting venlafaxine XR speeds onset of antidepressant action.

SECONDARY OUTCOMES:
To determine if hydrocortisone pre-treatment augments venlafaxine XR response.

CONTACTS AND LOCATIONS:
Overall Officials: Charles DeBattista, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States